CLINICAL TRIAL: NCT04410965
Title: Evaluation of the Relationship Between ABCG2 Mutation and Teriflunomide Exposure and Safety in Chinese RMS Patients Treated With Teriflunomide 14 mg Once Daily for 24 Weeks
Acronym: TERI-PK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDR16019; U1111-1233-0136 (Registry Identifier: ICTRP)
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- teriflunomide (Experimental): daily oral administration of teriflunomide 14 mg for 24 weeks
  Interventions: Drug: TERIFLUNOMIDE

INTERVENTIONS:
Drug: TERIFLUNOMIDE — Pharmaceutical form:tablet Route of administration: oral

SUMMARY:
Primary Objective:

Evaluate the relationship between ABCG2 mutation (rs2231142) and teriflunomide exposure, during 6-month treatment with teriflunomide 14 mg

Secondary Objective:

Characterize the safety (AEs, such as ALT enhancement, hair thinning, diarrhea, nausea, etc.) during 6-month treatment with teriflunomide

DETAILED DESCRIPTION:
Study duration per participant is approximately 28 weeks including a 24-week treatment period

ELIGIBILITY:
Inclusion criteria:

Participants are eligible to be included in the study only if all the following criteria apply:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Participants EDSS score ≤ 5.5 according to the diagnosis of the neurologist (using the 2017 Revised McDonald Diagnostic Criteria for MS) and upon treatment initiation with teriflunomide according to the approved product information in China.
* Participants will be genotyped for the rs2231142 mutation, enrolled 80 participants should include: 40 wildtype patients, 40 patients with ABCG2 (rs2231142) mutation
* Male and/or female participants:

  * Male participants: A male participant must agree to use contraception during the intervention period and undergo the accelerated eliminated procedure after the last dose of study intervention and refrain from donating sperm during this period.
  * Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance during the intervention period and undergo the accelerated elimination procedure (if necessary) after the last dose of study intervention.
* Participants who has signed written informed consent prior to entering the screening phase of the study

Exclusion criteria:

Participants are excluded from the study if any of the following criteria apply:

* Participant not willing /being able to complete the questionnaires and examination.
* Participants who have taken leflunomide within 2 years prior to screening.
* Participants who have taken teriflunomide within 2 years prior to screening.
* Participants with severe hepatic impairment, including active hepatitis B/C diagnosed.
* Known history of active tuberculosis (TB) or latent TB infection not adequately treated, either diagnosed by standard medical practice or guidelines.
* Relapse within 30 days prior to enrollment.
* Participants who have any contraindications to AUBAGIO according to the local product insert leaflet.
* History of a hypersensitivity of teriflunomide, leflunomide, or any the inactive ingredients in Aubagio.
* Human immunodeficiency virus (HIV) positive patients.
* Participants treated with:

  * glatiramer acetate, interferons, or dimethyl fumarate within 1 month prior to enrollment.
  * fingolimod, or intravenous immunoglobulins within 3 months prior to enrollment.
  * natalizumab, other immunosuppressant or immunomodulatory agents, such as cyclophosphamide, azathioprine, cyclosporine, methotrexate, mycophenolate, within 24 weeks prior to enrollment.
  * cladribine or mitoxantrone within 2 years prior to enrollment.
  * adrenocorticotrophic hormone (ACTH) or systemic corticosteroids for 2 weeks prior to enrollment.
* Participant treated with BCRP inhibitors (such as cyclosporine, eltrombopag, gefitinib).
* Participant not suitable for participation, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures.
* Any specific situation during study implementation/course that may rise ethics considerations.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
PK exposure: Cmax | From Week 8 to Week 24
  PK exposure Cmax will be estimated by PopPK analysis.
PK exposure: AUCtau | From Week 8 to Week 24
  PK exposure AUCtau will be estimated by PopPK analysis

SECONDARY OUTCOMES:
Participants with Serious Adverse Events and Adverse Events | Screening to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number, China, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Quan C, Zhou H, Yang H, Jiao Z, Zhang M, Zhang B, Tan G, Bu B, Jin T, Li C, Xue Q, Dong H, Shi F, Qin X, Zhang X, Gao F, Zhang H, Wang J, Hu X, Chen Y, Liu J, Qiu W. Safety of teriflunomide in Chinese adult patients with relapsing multiple sclerosis: A phase IV, 24-week multicenter study. Chin Med J (Engl). 2025 Feb 20;138(4):452-458. doi: 10.1097/CM9.0000000000002990. Epub 2024 Feb 5. PMID 38311806
- See also: BDR16019 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25217&tenant=MT_SNY_9011